CLINICAL TRIAL: NCT03746717
Title: Use of an Occlusive Skin Closure System May Reduce Post-operative Wound Drainage After Tumor Arthroplasty of the Hip
Brief Title: Occlusive Skin Closure May Reduce Wound Drainage After Tumor Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Werner Hettwer, Consultant Orthopaedic Oncology Surgeon, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRINEO-RCT RH-MSKTS-ORTH
Record Dates: First submitted 2018-11-04; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Bone Disease of the Proximal Femur

STUDY DESIGN:
Intervention Model Description: Open 2-arm prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prineo (Experimental): Skin closure with Dermabond Prineo occlusive wound closure system
  Interventions: Device: occlusive wound closure
- Staples (Active Comparator): Skin closure with staples
  Interventions: Device: conventional wound closure

INTERVENTIONS:
Device: occlusive wound closure — skin closure with a commercially available wound closure product consisting of a synthetic adhesive mesh and cyanoacrylate based skin glue
  Arms: Prineo
Device: conventional wound closure — wound closure with surgical staples
  Arms: Staples

SUMMARY:
Study Type: Investigator initiated, non-significant risk

Study Objective(s): To establish the effect of occlusive wound closure with the DERMABONDTM PRINEO skin closure system, compared to routine wound closure with skin staples, on post-operative wound discharge (PWD) after tumor arthroplasty of the hip

Study Population: Patients with secondary tumors of bone, undergoing tumor resection and primary endoprosthetic reconstruction involving the hip joint

Inclusion Criteria:

* Bone resection and endoprosthetic reconstruction for metastatic bone lesions involving the proximal femur or acetabulum
* Imminent, or de-facto pathologic fractures of proximal femur and/or acetabulum, requiring endoprosthetic reconstruction (with or without bone resection) involving the hip joint

Exclusion Criteria:

* Minors
* Pregnant and breast-feeding women
* Skin defects and wound conditions not amenable to primary wound closure and other DERMABOND PRINEO contraindications
* Underlying infection
* Total femur replacements
* Implant revision procedures

Structure: Open 2-arm prospective randomized controlled trial.

Duration of Study: 18 -24 months Multi-center: No Masking/Blinding: No Method of Subject Assignment: Block Randomization (10 in each block) Concurrent Control: Active - wound closure with skin staples Estimated Total Sample Size: 70 subjects will be enrolled in this study Statistical Rationale Provided: Yes Statistical Methods: Student t test for unpaired data

Study Endpoints:

* Time to dry wound status (in post-operative days)
* Duration of antibiotic use (in post-operative days)
* Length of hospital stay (in post-operative days)

DETAILED DESCRIPTION:
Background:

Patients undergoing bone tumor resection and subsequent endoprosthetic reconstruction are at significant risk of developing prosthetic joint infection (PJI)Additionally, numerous factors contribute to a significant predisposition of these patients to wound healing complications, including the burden of their primary disease, associated comorbidities, previous or ongoing treatment often involving chemotherapy and or radiotherapy, and the extent of the necessary surgical procedure. In a retrospective review of this specific patient population treated at the investigators institution during recent years, the investigators have found a very high prevalence of persistent discharge from the surgical wound, when routine wound closure with skin staples was used. This is of particular concern, as an association of this post-operative complication with a higher incidence of PJI has been clearly established in several large studies on conventional total hip arthroplasty. Another previous study showed that prolonged wound discharge (PWD) will often lead to increased length of hospital stay and increased use of antibiotics to prevent infection. In the same study, the investigators were able to demonstrate a substantial reduction of PWD, use of intra-venous antibiotics and length of hospital stay, with use of an alternative skin closure method, combining intradermal suture and Steristrips for optimal wound edge apposition and a topical skin adhesive (2-octyl cyanoacrylate) as a sealant. However, more extensive data on the prevalence of persistent surgical wound discharge and the preventive effect of skin adhesives as an adjunct to wound closure in high-risk patient populations are lacking in the literature.

Investigational Product:

The DERMABOND PRINEO Skin Closure System has been specifically developed with the goal to achieve fast and secure closure of long incisions. It consists of two components, a pressure sensitive adhesive (PSA) initiated flexible mesh, designed for wound edge approximation and a cyanoacrylate based topical skin adhesive for occlusive wound closure. Intradermal suture is not necessary, as this system has been shown to support wound closure strength equivalent to subcuticular 3-0 sutures and is able to provide even distribution of tension across the entire incision length to ensure wound edge approximation throughout the wound healing process. Furthermore, compared to subcuticular suture, it has demonstrated equivalent wound healing and cosmesis at 90 days, while reducing wound closure time by up to 70%. It also provides an immediately effective occlusive barrier with documented antimicrobial properties, enabling patients to shower directly following a procedure and can be easily removed after the patient's natural wound healing process is complete, estimated at anywhere between 12 to 25 days.

Aims of this study:

The investigators aim to evaluate wound closure with the DERMABOND PRINEO Skin Closure System in comparison to conventional wound closure with staples in 70 patients undergoing endoprosthetic joint replacement surgery for a metastatic bone tumor, involving the proximal femur or acetabular region, in a prospective randomized study and hypothesize that:

1. Skin closure with the DERMABOND PRINEO Skin Closure System will lead to a decreased PWD during the early post operative period.
2. Skin closure with the DERMABOND PRINEO Skin Closure System will lead to a decreased use of antibiotics during the early post operative period.
3. Skin closure with the DERMABOND PRINEO Skin Closure System will lead to shorter hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Bone resection and endoprosthetic reconstruction for metastatic tumors of the proximal femur or acetabulum
* Imminent, or de-facto pathologic fractures of proximal femur and/or acetabulum, requiring endoprosthetic reconstruction (with or without bone resection) involving the hip joint

Exclusion Criteria:

* Minors
* Pregnant and breast-feeding women
* Skin defects and wound conditions not amenable to primary wound closure and other DERMABONDTM PRINEOTM contraindications (see 5.1.3.)
* Underlying infection
* Total femur replacements
* Implant revision procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-11-03 (Actual)

PRIMARY OUTCOMES:
Wound status | Up to hospital discharge (approximately 1-2 weeks) measured in number of days from intervention
  time to dry wound status

SECONDARY OUTCOMES:
Antibiotic Use | Up to hospital discharge (approximately 1-2 weeks) measured in number of days from intervention
  time during which prophylactic antibiotics are administered

OTHER OUTCOMES:
Hospital Stay | Up to hospital discharge (approximately 1-2 weeks) measured in number of days from intervention
  time to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Werner H Hettwer, MD, MSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
It is not planned to share IPD